CLINICAL TRIAL: NCT00541775
Title: A Multicenter, Double-Blind, Placebo and Active Controlled, Randomized Study to Evaluate the Safety and Efficacy of the Addition of Sitagliptin 100 mg Once Daily in Patients With Type 2 Diabetes With Inadequate Glycemic Control on Metformin Monotherapy
Brief Title: Safety/Efficacy of Sitagliptin in Patient w/ Type 2 Diabetes (0431-801)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-801; 2007_623
Record Dates: First submitted 2007-10-05; First posted 2007-10-10 (Estimated); Results first posted 2010-06-17 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Sitagliptin (Experimental): sitagliptin 100 mg
  Interventions: Drug: Sitagliptin; Drug: Comparator: Metformin
- Rosiglitazone (Active Comparator): rosiglitazone 8 mg
  Interventions: Drug: Comparator: Rosiglitazone; Drug: Comparator: Metformin
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo; Drug: Comparator: Metformin

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg administered as one oral tablet once daily in the morning for up to 18 weeks.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Comparator: Rosiglitazone — Rosiglitazone 8 mg administered as two 4 mg capsules once daily in the morning for up to 18 weeks.
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Comparator: Placebo — placebo - administered as one placebo tablet to match Sitagliptin 100 mg and two placebo capsules to match rosiglitazone 4 mg once daily in the morning for up to 18 weeks.
  Arms: Placebo
Drug: Comparator: Metformin — Open-label metformin was supplied by the Sponsor as 500, 850, or 1000 mg oral tablets administered at a daily dose of >= 1500 mg.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of sitagliptin in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patient has Type 2 diabetes
* Currently taking metformin >1500 mg/day for at least 10 weeks
* Male or female

Exclusion Criteria:

* Patient has peripheral edema
* History of type 1 diabetes
* Patient required insulin within prior 8 weeks
* Have participated or are currently participating in another study with an investigational compound or device within 12 weeks of starting this study
* Participating in a weight loss program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2006-06; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Scott R, Loeys T, Davies MJ, Engel SS; Sitagliptin Study 801 Group. Efficacy and safety of sitagliptin when added to ongoing metformin therapy in patients with type 2 diabetes. Diabetes Obes Metab. 2008 Sep;10(10):959-69. doi: 10.1111/j.1463-1326.2007.00839.x. Epub 2008 Jan 14. PMID 18201203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 16-June-2006. Last Patient Last Visit: 2-March-2007. 13 medical clinics in 3 countries in Europe and 23 in 4 countries in the rest of the world
Pre-assignment Details: Patients 18-75 years of age with type 2 diabetes mellitus (T2DM) who were taking metformin monotherapy at a stable dose of ≥ 1500 mg/day for at least 10 weeks and had inadequate glycemic control (hemoglobin A1C ≥ 7.0% and ≤11%) were eligible to participate.
Groups:
- Sitagliptin: The Sitagliptin group includes data from patients randomized to receive treatment with oral tablets of sitagliptin 100 mg and placebo matching rosiglitazone q.d. (once-daily) with metformin (≥1500 mg/day).
- Rosiglitazone: The Rosiglitazone group includes data from patients randomized to receive treatment with oral tablets of rosiglitazone 8 mg and placebo matching sitagliptin q.d. in combination with metformin (≥1500 mg/day).
- Placebo: The Placebo group includes data from patients randomized to receive treatment with oral tablets of placebo matching sitagliptin and placebo matching rosiglitazone q.d. with metformin (≥1500 mg/day).
Period: Overall Study
Arm/Group | Sitagliptin | Rosiglitazone | Placebo
Started | 94 | 87 | 92
Completed | 85 | 85 | 84
Not Completed | 9 | 2 | 8
Not completed — Adverse Event | 3 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject and Other | 5 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Rosiglitazone | Placebo | Total
Number analyzed (Participants) | 94 | 87 | 92 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.8) | 54.8 (10.5) | 55.3 (9.3) | 55.1 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 32 | 38 | 112
  Male | 52 | 55 | 54 | 161
Race/Ethnicity, Customized [Number; unit: participants]
  White | 57 | 51 | 56 | 164
  Black | 0 | 1 | 0 | 1
  Asian | 36 | 33 | 36 | 105
  Other | 1 | 2 | 0 | 3
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 157.5 (31.4) | 156.9 (31.6) | 160.0 (37.4) | 158.1 (33.5)
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin (A1C)] | 7.8 (1.0) | 7.7 (0.8) | 7.7 (0.9) | 7.7 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C (A1C) at Week 18
Description: A1C is measured as percent. Thus, this change from baseline reflects the Week 18 A1C percent minus the Week 0 A1C percent.
  The study hypothesis comparison was between sitagliptin versus placebo.
Time Frame: Baseline and 18 Weeks
Population: The all patients treated population included all patients who took at least one dose of study medication and had both a baseline measurement and at least one post-randomization measurement for this outcome. Missing data were imputed using the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin (A1C)
Arm/Group | Sitagliptin | Rosiglitazone | Placebo
Number analyzed (Participants) | 91 | 87 | 88
Percent of glycosylated hemoglobin (A1C) | -0.73 [-0.87 to -0.60] | -0.79 [-0.92 to -0.65] | -0.22 [-0.36 to -0.08]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p <= 0.001, ANCOVA; Analysis of covariance with a term for treatment, and a covariate for baseline value; Mean Difference (Net) = -0.51, 95% CI [-0.70 to -0.32], Standard Error of Mean 0.1

2. Secondary Outcome: Fasting Plasma Glucose (FPG) at Week 18
Description: The change from baseline is the Week 18 FPG minus the Week 0 FPG.
Time Frame: Baseline and 18 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Rosiglitazone | Placebo
Number analyzed (Participants) | 92 | 87 | 89
mg/dL | -11.7 [-18.6 to -4.9] | -24.5 [-31.6 to -17.5] | 6.1 [-0.8 to 13.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p <= 0.001, ANCOVA; Analysis of covariance with a term for treatment, and a covariate for baseline value; Mean Difference (Net) = -17.8, 95% CI [-27.6 to -8.1], Standard Error of Mean 5

3. Secondary Outcome: 2-hour Post-meal Glucose (PMG) at Week 18
Description: The change from baseline is the Week 18 PMG minus the Week 0 PMG.
Time Frame: Baseline and 18 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Rosiglitazone | Placebo
Number analyzed (Participants) | 80 | 76 | 78
mg/dL | -35.4 [-46.3 to -24.5] | -51.3 [-62.5 to -40.1] | -4.9 [-16.0 to 6.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority or Other; p <= 0.001, ANCOVA; Analysis of covariance with a term for treatment, and a covariate for baseline value; Mean Difference (Net) = -30.5, 95% CI [-46.0 to -15.0], Standard Error of Mean 7.9

ADVERSE EVENTS:
Time Frame: Weeks 0 to 18
Description: Safety tables are based on the All Patients as Treated (APaT) population that includes all patients who took at least one dose of study drug. One patient in the placebo group did not take any study drug. Thus, for the placebo group 92 patients are reported in the baseline characteristics and 91 patients are reported in the AE summary.
Arm/Group | Sitagliptin | Rosiglitazone | Placebo
Serious Adverse Events (participants affected / at risk) | 5/94 | 5/87 | 5/91
Other Adverse Events (participants affected / at risk) | 5/94 | 1/87 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=94) | Rosiglitazone (N=87) | Placebo (N=91)
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 3 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin (N=94) | Rosiglitazone (N=87) | Placebo (N=91)
Blood glucose increased (Investigations) | 5 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.